CLINICAL TRIAL: NCT06611904
Title: Study of Endothelial Glycocalyx and Vascular Function in Patients With Type 2 Diabetes and Albuminuria After Administration of Dulaglutide and Dapagliflozin vs DPP-4 Inhibitors
Brief Title: The Effect of Combined Dulaglutide and Dapagliflozin Treatment vs DPP-4 Inhibitors in Endothelial and Vascular Function in Patients With Type 2 Diabetes Mellitus and Albuminuria
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine and Endocrinology, Attikon Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 456/11-06-2017
Record Dates: First submitted 2024-09-20; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Urine Albumin (UAlb); Glycocalyx; Arterial Stiffness
Keywords: type 2 diabetes; albuminuria; arterial stiffness; glycocalyx
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Albuminuria | interventions — dulaglutide; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving dulaglutide and dapagliflozin (Active Comparator): Patients with T2DM and albuminuria receiving dulaglutide and dapagliflozin
  Interventions: Drug: Dulaglutide
- Patients receiving DPP-4i (Active Comparator): Patients with T2DM and albuminuria receiving DPP-4i
  Interventions: Drug: DPP-4 Inhibitors

INTERVENTIONS:
Drug: Dulaglutide — Combined treatment with dulaglutide and dapagliflozin
  Arms: Patients receiving dulaglutide and dapagliflozin
Drug: DPP-4 Inhibitors — DPP-4i treatment as an add-on to metformin
  Arms: Patients receiving DPP-4i

SUMMARY:
Patients with Type 2 Diabetes Mellitus and albuminuria will be randomised eitheer to dulaglutide and dapagliflozin combination or DPP-4 inhibitor, as an add-on treatment to metformin. Arterial stiffness, UACR, endothelial glycocalyx and global longitudinal strain will be assesed at baseline, 4 and 12 months.

DETAILED DESCRIPTION:
Patients with Type 2 Diabetes Mellitus and albuminuria will be randomised eitheer to dulaglutide and dapagliflozin combination or DPP-4 inhibitor, as an add-on treatment to metformin. Arterial stiffness via pulse wave velocity (PWV), UACR, endothelial glycocalyx via Microscan camera, and global longitudinal strain via echocardiography will be assesed at baseline, 4 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus Albuminuria HbA1c: 7-10% eGFR> 60 ml/min

Exclusion Criteria:

* Type 1 diabetes mellitus Inflammation, chronic or acute Established cardiovascular disease Malignancy within the last 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
UACR | 4 and 12 months
  UACR change after 4 and 12 months of treatment
PWV | 4 and 12 months
  PWV change after 4 and 12 months of treatment
PBR | 4 and 12 months
  PBR change after 4 and 12 months of treatment
GLS | 4 and 12 months
  GLS change after 4 and 12 months of ttreatment

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University General Hospital, Chaïdári, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lambadiari V, Pavlidis G, Kousathana F, Maratou E, Georgiou D, Andreadou I, Kountouri A, Varoudi M, Balampanis K, Parissis J, Triantafyllidi H, Katogiannis K, Birba D, Lekakis J, Dimitriadis G, Ikonomidis I. Effects of Different Antidiabetic Medications on Endothelial Glycocalyx, Myocardial Function, and Vascular Function in Type 2 Diabetic Patients: One Year Follow-Up Study. J Clin Med. 2019 Jul 5;8(7):983. doi: 10.3390/jcm8070983. PMID 31284526
- [Result] Lambadiari V, Pavlidis G, Kousathana F, Varoudi M, Vlastos D, Maratou E, Georgiou D, Andreadou I, Parissis J, Triantafyllidi H, Lekakis J, Iliodromitis E, Dimitriadis G, Ikonomidis I. Effects of 6-month treatment with the glucagon like peptide-1 analogue liraglutide on arterial stiffness, left ventricular myocardial deformation and oxidative stress in subjects with newly diagnosed type 2 diabetes. Cardiovasc Diabetol. 2018 Jan 8;17(1):8. doi: 10.1186/s12933-017-0646-z. PMID 29310645
- [Derived] Korakas E, Thymis J, Oikonomou E, Mourouzis K, Kountouri A, Pliouta L, Pililis S, Pavlidis G, Lampsas S, Katogiannis K, Palaiodimou L, Tsivgoulis G, Siasos G, Ikonomidis I, Raptis A, Lambadiari V. Dulaglutide and Dapagliflozin Combination Concurrently Improves the Endothelial Glycocalyx and Vascular and Myocardial Function in Patients with T2DM and Albuminuria vs. DPP-4i. J Clin Med. 2024 Dec 10;13(24):7497. doi: 10.3390/jcm13247497. PMID 39768420